CLINICAL TRIAL: NCT03425201
Title: A Phase I-II Study to Evaluate the Efficacy and Safety of Niraparib in Combination with Cabozantinib (XL184) in Patients with Advanced Urothelial Cancer After Failure to First-line Platinum-based Chemotherapy
Brief Title: Niraparib in Combination with Cabozantinib (XL184) in Patients with Advanced Urothelial Cancer (NICARAGUA)
Acronym: NICARAGUA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundacion CRIS de Investigación para Vencer el Cáncer (Other)
Collaborators: Ipsen (Industry); GlaxoSmithKline (Industry); Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NICARAGUA; 2017-004367-12 (EudraCT Number)
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Urothelial Cancer
MeSH Terms: interventions — niraparib; cabozantinib

STUDY DESIGN:
Intervention Model Description: Open-label, multicenter, phase I/II dose-escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Niraparib plus Cabozantinib (Experimental): Patients will receive niraparib and cabozantinib p.o. once daily in 28-day cycles.
  In phase I, patients will be accrued to each dose level in cohorts of 6 patients. Escalation will continue until a dose-limiting toxicity (DLT) is observed or the highest dose-level is reached.
  In phase II study patients will receive niraparib p.o. once daily and cabozantinib p.o. once daily in 28-day cycles at doses recommended in the phase I study.
  If niraparib or cabozantinib need to be interrupted due to toxicity, patient can continue only with the other drug.
  Interventions: Drug: Niraparib plus Cabozantinib

INTERVENTIONS:
Drug: Niraparib plus Cabozantinib — Non-randomized trial will comprise 2 stages. A dose escalation phase will characterize the safety, tolerability, DLTs and MTD, of oral niraparib plus cabozantinib in patients with urothelial or renal cell carcinoma. Subsequently, the phase II will further evaluate the safety and antitumor activity of this combination in patients with urothelial carcinoma.

SUMMARY:
Cabozantinib is an oral, small-molecule tyrosine kinase inhibitor. Its primary targets are Hepatocyte growth factor receptor protein (MET), vascular endothelial growth factor receptor 1-3 (VEGFR1-3), RET, AXL, FLT3 and KIT. Cabozantinib has been approved by the FDA for clinical treatment of progressive, metastatic medullary thyroid cancer. Recently published trials have demonstrated activity for cabozantinib in patients with advanced renal cell carcinoma and metastatic castration-resistant prostate cancer (mCRPC). Furthermore, in preclinical models of urothelial carcinoma (UC) of the bladder, cabozantinib has demonstrated the ability to inhibit tumor xenograft growth. It has been suggested that levels of soluble Met ectodomain (sMet) can be measured in the urine as a useful biomarker to monitor the efficacy of c-Met therapy in bladder cancer patients. Moreover, cabozantinib has demonstrated activity in heavily pretreated, advanced bladder cancer patients, with a response rate of 19.5% and manageable toxicities.

In the phase I of this study it is proposed to evaluate DLTs of niraparib and cabozantinib combination and determine maximum tolerated dose (MTD) in patients with advanced urothelial or renal cell carcinoma. In the phase II it is proposed to make a preliminary evaluation of the efficacy of this combination in patients with urothelial cell carcinoma. Efficacy results will be correlated with genomic alterations related to c-Met and Poly [ADP-ribose] polymerase (PARP) inhibitor activity.

DETAILED DESCRIPTION:
Bladder cancer is the 9th most common cancer worldwide, with around 429.800 new cases diagnosed in 2012 and the 5th most common cancer in Europe, with more than 151.000 new cases diagnosed in 2012. Relating mortality figures, bladder cancer is the 13th most common cause of cancer death worldwide, with around 165.100 deaths from bladder cancer in 2012 and the 9th in Europe, with around 52.400.

Cisplatin-based chemotherapy remains the standard treatment in patients with metastatic urothelial carcinoma (UC).This regimen has been associated with a median survival of 14-15 months. The prognosis of patients who progress after a platinum-based regimen is dismal. Several chemotherapy drugs tested in the second-line setting, such as taxanes, vinflunine and pemetrexed, have demonstrated limited activity, with response rates of 5-20%, median progression-free survival (PFS) of 2-4 months, and median survival of 6-8 months. Thus, there are significant unmet medical needs in the second-line setting. New therapeutic targets should be tested in urothelial carcinoma to improve these results.

Therapies targeting DNA repair pathways can exploit DNA repair defects in cancer cells to generate synthetic lethality. Alterations in DNA repair pathways have been associated with response to DNA-damaging agents. For example, defective homologous recombination (HR) plays a crucial role in tumors where platinum agents are involved in therapeutic management, as well as in those treated with PARP inhibitors, which have synthetic lethal effects when applied to cells with defective HR. Targeted mutational profiling of HR genes using next-generation sequencing has been used to identify mutations of key HR genes. Furthermore, HR-defective tumors exhibit genomic instability, including loss of heterozygosity (LOH), telomeric allelic imbalance (TAI) and large-scale state transitions (LST). A combined HR deficiency score (myChoice homologous recombination deficiency (HRD) test from Myriad Genetics) defined as the sum of LOH, TAI and LST has been developed. This score has been associated with response to platinum-based chemotherapy and in ovarian cancer with the efficacy of niraparib in patients without germline breast cancer gene (gBRCA) mutations.

In patients with muscle-invasive bladder cancer (MIBC), the Cancer Genome Atlas project found 31% of alterations in BRCA1-2 genes, mainly related to copy number and overexpression. In addition, a high percentage of tumors had alterations in other DNA repair genes. Recently, in platinum-treated UC patients, 47% of mutations in DNA repair genes have been found, including 50% of mutations in HR, Fanconi anemia, and DNA-damage-response checkpoint pathways. The presence of these mutations has been associated with survival. These results suggest a potential role for PARP inhibitors in UC. Niraparib is a highly selective inhibitor of poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP)1/2 nuclear protein. PARP enzymes are involved in DNA repair through activation of the base excision repair (BER) pathway and alternative end-joining pathways and inhibition of non-homologous end-joining. PARP inhibition in cells with HR deficiency causes accumulation of unrepaired DNA double-strand breaks, leading to cell death. For these reasons, PARP inhibitors are selectively lethal in tumor cells with defective HR. Niraparib at the recommended oral dose of 300 mg daily has demonstrated efficacy in platinum- sensitive recurrent ovarian cancer with defective HR. The most significant toxicity was hematologic (thrombocytopenia, neutropenia, and anemia). Among non-hematologic toxicities, hypertension was detected in 8% of patients.

c-Met receptor tyrosine kinase (RTK) is activated by its ligand, hepatocyte growth factor (HGF), and induces increased proliferation, migration, motility, and invasion of bladder cancer cells. c-Met is overexpressed in more than 60% of metastatic bladder cancer patients and is linked to poor outcome. Furthermore, in bladder cancer, c-Met is co-expressed with other RTKs, such as AXL and PDGFR. Some evidence suggests a relationship between c-Met and AXL expression with DNA damage response and resistance to chemotherapy. For example, Balaji et al have demonstrated that AXL inhibition leads to a defect in the HR pathway, sensitizing cells to PARP inhibition. In a recently published study, a significant interaction between c-Met and Poly [ADP-ribose] polymerase 1 (PARP1) was detected in breast cancer cell lines. c-Met activity can decrease response to PARP inhibitors, whereas treatment with c-Met inhibitors renders cells more sensitive to PARP inhibition. Likewise, in in vivo models with xenograft tumors, the combination of c-Met and PARP inhibitors showed a significant reduction in tumor growth compared to either inhibitor alone. This interaction can be explained because c-Met mediates PARP1 function through phosphorylation of PARP1 at Y907. These results raise the possibility that bladder cancer patients with tumors overexpressing c-Met can benefit from the combination of c-Met inhibitors and PARP inhibitors.

Cabozantinib is an oral, small-molecule tyrosine kinase inhibitor. Its primary targets are MET, VEGFR1-3, RET, AXL, FLT3 and KIT. Cabozantinib has been approved by the FDA for clinical treatment of progressive, metastatic medullary thyroid cancer. The recommended dose of cabozantinib has been established in phase I trials at 60 mg/day in 28-day cycles. Recently published trials have demonstrated activity for cabozantinib in patients with advanced renal cell carcinoma and metastatic castration-resistant prostate cancer (mCRPC). Furthermore, in preclinical models of UC of the bladder, cabozantinib has demonstrated the ability to inhibit tumor xenograft growth. It has been suggested that levels of soluble Met ectodomain (sMet) can be measured in the urine as a useful biomarker to monitor the efficacy of c-Met therapy in bladder cancer patients. Moreover, cabozantinib has demonstrated activity in heavily pretreated, advanced bladder cancer patients, with a response rate of 19.5% and manageable toxicities.

In the phase I of this study it is proposed to evaluate DLTs of niraparib and cabozantinib combination and determine MTD in patients with advanced urothelial or renal cell carcinoma. In the phase II it is proposed to make a preliminary evaluation of the efficacy of this combination in patients with urothelial cell carcinoma. Efficacy results will be correlated with genomic alterations related to c-Met and PARP inhibitor activity.

ELIGIBILITY:
Inclusion Criteria:

Phase I study:

1. Histologically confirmed UC of the urinary tract or renal cell carcinoma
2. Advanced or metastatic disease that is not amenable to curative surgery or radiation
3. Patients must be willing to provide a tumor specimen prior to enrollment
4. Previous therapy:

   i.Renal cell carcinoma: Prior tyrosine kinase inhibitor (TKI) and mechanistic target of rapamycin (mTOR) therapies is allowed ii.UC of the urinary tract: ≤2 previous chemotherapy regimens (including a platinum-based regimen)
5. Measurable disease will not be required
6. The remaining inclusion/exclusion criteria will be identical to the phase II study
7. Recovery to at least grade I from toxicities related to prior treatment unless non clinically significant or stable on supportive therapy

Phase II study:

1. Age ≥18 years
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤1
3. Histologically confirmed UC of the bladder, urethra, ureter or renal pelvis (patients with mixed histologies will be allowed if urothelial is the predominant component).
4. Patients must have formalin-fixed paraffin-embedded (FFPE) tumor samples available from the primary or recurrent cancer or agree to undergo fresh biopsy prior to study treatment initiation
5. Advanced or metastatic disease that is not amenable to curative surgery or radiation
6. Prior treatment with one prior cytotoxic regimen of platinum-based chemotherapy. If the only prior cytotoxic therapy was administered in perioperative (ie, neoadjuvant or adjuvant) settings, the patient will be eligible provided the interval from end of therapy to the diagnosis of metastatic disease is less than one year.
7. Confirmed progressive disease after treatment with platinum-based chemotherapy
8. At least one measurable disease site that has not been previously irradiated
9. No prior therapy with Poly(ADP-ribose) polymerase (PARP) or c-Met inhibitors.
10. Prior anti programmed cell death protein 1 (PD1) and anti programmed death-ligand 1 (PD-L1) therapy is permitted
11. Adequate bone marrow, liver and renal functions as assessed by the following:

    * Hemoglobin ≥9 g/dL; absolute neutrophil count ≥1500 cells/µL; platelets ≥100,000 g/µL;
    * Total bilirubin ≤1.5 times upper limit of normal (ULN) (≤2.0 in patients with known Gilberts syndrome); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times ULN unless liver metastases are present, in which case they must be ≤5x ULN.
    * Serum creatinine ≤1.5x ULN or creatinine clearance ≥30 mL/min using Cockcroft-Gault formula
    * Urine protein/creatinine ratio (UPCR) ≤1 mg/mg (113.2 mg/mmol) creatinine or 24-hr urine protein of <1 g
12. Life expectancy greater than 3 months
13. Patients must be able to take oral medications
14. Participant receiving corticosteroids may continue as long as their dose is stable for least 4 weeks prior to initiating protocol therapy.
15. Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
16. Female participant has a negative serum pregnancy test within 7 days prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study treatment, or is of non-childbearing potential. Non-childbearing potential is defined as follows (by other than medical reasons):

    * ≥45 years of age and has not had menses for >1 year
    * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation a. Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 180 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
17. Participant must agree to not breastfeed during the study or for 180 days after the last dose of study treatment.
18. Male participant agrees to use an adequate method of contraception starting with the first dose of study treatment through 180 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
19. Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent

Exclusion Criteria:

1. Participant must not be simultaneously enrolled in any interventional clinical trial
2. Major surgery, open biopsy or significant traumatic injury within 8 weeks prior to study entry and complete wound healing at the inclusion
3. Participant must not have received investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior initiating protocol therapy.
4. Progressed while on platinum treatment or within 2 months from completion of platinum-containing regimen. Exclusion criteria applicable only to patients included in phase II.
5. Radiation therapy for bone or brain metastases within 4 weeks before first dose of study drug. Other external radiation within 4 weeks before first dose of study drug. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible
6. Participant must not have a known hypersensitivity to niraparib or cabozantinib components or excipients.
7. Participant must not have received a transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy.
8. Participant must not have received colony stimulating factors (eg, granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy.
9. Participant has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
10. Known history of myelodysplastic syndrome (MDS) or a pre-treatment cytogenetic testing result at risk for a diagnosis of MDS/acute myeloid leukemia (AML)
11. Unstable systemic disease or active uncontrolled infection
12. Any concurrent active malignancy requiring treatment (other than basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or malignancies curatively treated > 3 years prior to study entry)
13. Known uncontrolled symptomatic brain or leptomeningeal metastases or cranial epidural disease; subjects with brain metastases previously treated and on stable dose of corticosteroids and/or anticonvulsants for >4 weeks, or not requiring such medications, are eligible. Baseline brain scans are not required to confirm eligibility.
14. Uncontrolled hypertension
15. Significant cardiovascular diseases, clinically relevant cardiac arrhythmia, unstable angina or myocardial infarction within 6 months prior to randomization, congestive heart failure > New York Heart Association (NYHA) III, severe peripheral vascular disease, QT prolongation >470 msec ,clinically significant pericardial effusion
16. Receiving concomitant medications that prolong corrected QT and is unable to discontinue use
17. Concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or Factor Xa inhibitors, or antiplatelet agents (eg, clopidogrel). Low dose aspirin (≤ 100 mg/day), low-dose warfarin (≤ 1 mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted
18. Prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) test ≥1.3 x ULN within 7 days before the first dose of study treatment
19. Significant thromboembolic or vascular disorders within 6 months prior to administration of study drugs, including:

    * Symptomatic pulmonary embolism
    * Cerebrovascular accident
    * Peripheral arterial ischemia > grade 2
    * Coronary or peripheral artery bypass graft
20. The subject has experienced any of the following within 3 months before the first dose of study treatment:

    * clinically significant hematemesis or gastrointestinal bleeding
    * clinically significant hemoptysis
21. Any malabsorption problem that, in the investigator's opinion, would prevent adequate absorption of the study drug
22. Patient has not recovered to baseline or CTCAE ≤ Grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant Adverse Events
23. History of organ transplant
24. Concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment
25. Active infection requiring systemic treatment within 28 days before the first dose of study treatment
26. Serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
27. Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

    * Any of the following within 28 days before the first dose of study treatment: intra-abdominal tumor/metastases invading gastrointestinal mucosa, active peptic ulcer disease,inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
    * Any of the following within 6 months before the first dose of study treatment: History of abdominal fistula, gastrointestinal perforation, bowel obstruction or gastric outlet obstruction or intra-abdominal abscess
28. Chronic concomitant treatment of strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's Wort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Phase I: maximum tolerated dose | up to 1 month
  Highest dose at which ≤1 out of 6 patients experience a DLT
Phase II: progression free survival | Up to 6 months
  Time from the date of first dose of study treatment to the date of progression or death (from any cause).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 6 months
  Number of events per patient
Phase II: Objective Response Rate | Up to 6 months
  Response according to RECIST 1.1 criteria
Phase II: Disease Control Rate | Up to 6 months
  Response according to RECIST 1.1 criteria
Phase II: Duration of response | Up to 6 months
  Time from the date of response is achieved until documented tumor progression
Phase II: Overall Survival | Up to 6 months
  Time from the date of first dose of study treatment to the date of death due to any cause

OTHER OUTCOMES:
Correlation of the activity of niraparib plus cabozantinib with the molecular profile of the tumor | Up to 6 months
  Immunohistochemistry and RNA analysis of pre- and post-tumor samples

CONTACTS AND LOCATIONS:
Overall Officials: Albert Font, MD, Principal Investigator — ICO Badalona-Hospital Germans Trias i Pujol; Daniel Castellano, MD, Principal Investigator — Hospital 12 de Octubre
Locations (10):
- Spain (10):
  - Xarxa Assistencial Universitària de Manresa, Barcelona, Catalonia
  - ICO Badalona, Badalona
  - Hospital Clinic, Barcelona
  - ICO Girona, Girona
  - ICO L'Hospitalet, L'Hospitalet de Llobregat
  - Hospital 12 de Octubre, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Marques de Valdecilla, Santander
  - Instituto Valenciano de Oncología, Valencia

IPD SHARING:
Plan to Share IPD: No